CLINICAL TRIAL: NCT05133310
Title: Effect of Simvastatin on Sepsis and Febrile Neutropenia in Patients With Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Christian Omar Ramos-Peñafiel, MD, PhD, Principal Investigator, Hospital General de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGMDI/21/204/03/63
Record Dates: First submitted 2021-11-15; First posted 2021-11-24 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Strains; Acute Lymphoblastic Leukemia; Sepsis
Keywords: Acute lymphoblastic leukemia; Sepsis; Febrile Neutropenia; Simvastatin
MeSH Terms: conditions — Sprains and Strains; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Sepsis; Febrile Neutropenia | interventions — Simvastatin

STUDY DESIGN:
Intervention Model Description: Clinical randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care Group (No Intervention): Patients will receive the standard chemotherapy regimen assigned for their treatment and, they will be followed and monitored until the end of treatment and hospitalization.
- Simvastatin Treatment Group (Experimental): Patients will combine the standard CALGB treatment scheme plus Simvastatin 10mg orally every 24 hours during the first 7 days of treatment and then continue with 20mg every 24 hours until the end of treatment and hospitalization.
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Combination of Simvastatin with Standard Chemotherapy scheme for acute lymphoblastic patients.
  Other Names: Intervention Group
  Arms: Simvastatin Treatment Group

SUMMARY:
In general, the percentage of complete remissions is 85 - 90 % for acute lymphoid leukemia (ALL). In developing countries, percentages are lower secondary to higher sepsis-related mortality. Although the effect of statins on inflammatory response associated with sepsis has been demonstrated, including an effect on bacterial proliferation in patients with a state of immunosuppression, their effect has not been demonstrated so far in patients with hemato-oncological cancer.

DETAILED DESCRIPTION:
Death associated with sepsis is one of the principal complications related to chemotherapy treatment; there are currently no strategies to prevent its development besides the use of prophylactic antibiotics or granulocyte colony stimulants to reduce the period of febrile neutropenia. Most of the trials on the use of statins are retrospective with controversial results and include patients with different clinical situations that conditioned the septic study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute leukemia under treatment of a chemotherapy regimen
* Stable performance status (ECOG: 0 or Karnofsky scale greater than 80%) at time of analysis and under chemotherapy regimen
* Life expectancy greater than 48 hours after diagnosis
* Oral route available
* Have signed informed consent at the time of the study
* Patients whose chemotherapy regimen is administered in a hospital rather than an outpatient manner

Exclusion Criteria:

* Patients with acute leukemias over 55 years of age and with impaired functional status at the time of diagnosis
* Elevation of liver enzymes 3 times higher than the range established by the central laboratory
* Persistent kidney involvement despite having adequate hydration
* Pregnant patients
* Patients with peripheral neuropathy considered severe or disabling grade
* Patients with a history of psychiatric disorders or psychotic attacks
* Individuals who do not have the oral route available, who are maintained with a nasogastric tube, or who require support for the diagnosis through parenteral nutrition
* Patients undergoing peritoneal dialysis or hemodialysis treatment
* Patients with leukemia associated with Down syndrome
* Patients under low-intensity chemotherapy regimen or palliative regimen
* Previous allergy to any statin component
* Patients with a history of liver failure (Child-Pugh Stage B or C)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-12-16 (Estimated); Study Completion 2023-06-23 (Estimated)

PRIMARY OUTCOMES:
Hospital Discharge | 3 months
  The event in which patient is discharge from Hospital stay,
Feverish Event | 3 months
  Determination of a temperature above 38 ° persistently for more than 30 minutes
Sepsis | 3 months
  Presence of hemodynamic alterations characterized by persistent hypotension, elevated heart rate, fever, and abnormal respiration
Neutrophils count | 3 months
  Number of neutrophils found in peripheral blood at the end of each chemotherapy cycle
Platelets count | 3 month
  Number of platelets found in peripheral blood at the end of each chemotherapy cycle
Blasts in marrow | 3 month
  Presence of more than 5% of blasts in bone marrow after each chemotherapy cycle
Neutrophil recovery time | 1 month
  Time in days for neutrophil recovery

SECONDARY OUTCOMES:
Bacterial isolation | 3 months
  Description of the germ isolated in cultures during follow-up
Procalcitonin | 3 months
  Biomarker used in infectious and inflammatory processes associated mainly with gram-negative germs, this measurement is routine in the follow-up of individuals with febrile neutropenia
Hospital Stay | 1 month
  Measurement of days of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Martinez Tovar, PhD, Study Director — Hospital General de Mexico
Locations (1):
- Hospital General de México "Dr. Eduardo Liceaga", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
All participants and their information will be managed by intern investigators and will be kept secure for personal data protection according to Mexican laws.

REFERENCES:
- [Background] Escrihuela-Vidal F, Laporte J, Albasanz-Puig A, Gudiol C. Update on the management of febrile neutropenia in hematologic patients. Rev Esp Quimioter. 2019 Sep;32 Suppl 2(Suppl 2):55-58. PMID 31475812
- [Background] Pirzad Jahromi G, P Shabanzadeh A, Mokhtari Hashtjini M, Sadr SS, Rasouli Vani J, Raouf Sarshoori J, Charish J. Bone marrow-derived mesenchymal stem cell and simvastatin treatment leads to improved functional recovery and modified c-Fos expression levels in the brain following ischemic stroke. Iran J Basic Med Sci. 2018 Oct;21(10):1004-1012. doi: 10.22038/IJBMS.2018.29382.7100. PMID 30524673
- [Background] Pertzov B, Eliakim-Raz N, Atamna H, Trestioreanu AZ, Yahav D, Leibovici L. Hydroxymethylglutaryl-CoA reductase inhibitors (statins) for the treatment of sepsis in adults - A systematic review and meta-analysis. Clin Microbiol Infect. 2019 Mar;25(3):280-289. doi: 10.1016/j.cmi.2018.11.003. Epub 2018 Nov 23. PMID 30472427